CLINICAL TRIAL: NCT04011735
Title: A Real-world Non-interventional Study to Assess Patient Satisfaction With and Preference for Re-usable Respimat Soft Mist Inhaler in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Re-usable Respimat® Soft MistTM Inhaler Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0097
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol; tiotropium-olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Respimat SMI-experienced: Switching to re-usable Respimat: patients who had been on maintenance treatment with a disposable Respimat and who switched to a re-usable Respimat SMI at study entry.
  Interventions: Drug: Respimat
- Respimat SMI-naïve: patients who have not previously used a Respimat SMI product and receive their first prescription at study entry
  Interventions: Drug: Respimat
- Respimat SMI-experienced: Maintenance treatment: patients who have been on maintenance treatment with a Respimat SMI product and receive a refill prescription at study entry.

INTERVENTIONS:
Drug: Respimat — Soft Mist Inhaler product
  Other Names: (Spiriva®, Striverdi® or; Spiolto®)
  Groups: Respimat SMI-experienced: Switching to re-usable Respimat; Respimat SMI-naïve

SUMMARY:
The study is to assess patient satisfaction with the inhaler attributes of the re-usable Respimat SMI (Spiriva, Striverdi or Spiolto) in patients with COPD, including patients who are Respimat SMI-experienced and Respimat SMI-naïve. This study also aims to examine patient preference for the re-usable Respimat SMI compared to the disposable Respimat SMI in Respimat SMI-experienced patients switching from a disposable to a re-usable Respimat SMI product at study entry.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all the following inclusion criteria will be eligible for participation in the study:

* Provision of signed informed consent prior to study data collection
* Patient with COPD aged 40 years or older
* Patient prescribed (or already receiving the disposable Respimat SMI and switched to) one of the following re-usable Respimat SMI products per the standard clinical practice: Spiriva 2.5 microgram inhalation solution; (2) Striverdi 2.5 microgram inhalation solution; and (3) Spiolto 2.5 microgram / 2.5 microgram inhalation solution
* Patient unlikely to change their Respimat therapy during the 4-6 week observation period (in the opinion of the investigator)

Exclusion Criteria:

Patients fulfilling any of the following exclusion criteria will not be eligible for participation in the study:

* Patient using a disposable Respimat SMI product during the study period
* Patient who have had a severe COPD exacerbation requiring hospitalisation in the immediate 3 months prior to study entry
* Patient participating in a clinical trial or any other non-interventional study of a drug or device at the time of enrolment
* Visual, cognitive, motor or health impairment that, as judged by the investigator, may cause concern regarding the patient's ability to complete the questionnaires
* Patient not fluent and literate in one of the main languages of the country

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is planned that approximately with 250 Chronic Obstructive Pulmonary Disease (COPD) patients (Respimat SMI-experienced and Respimat SMI-naïve) from Europe will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Belgium (3):
  - Brussels - UNIV UZ Brussel, Brussels
  - Clinique Notre-Dame de Grâce, Gosselies
  - Roeselare - HOSP AZ Delta, Menen
- Denmark (2):
  - Hvidovre Hospital, Hvidovre
  - Vejle Hospital, Vejle
- TYKS, Keuhkosairauksien klinikka, Turku, Turku, Finland
- Germany (5):
  - Universitätsklinikum Aachen, AöR, Aachen
  - MECS Research GmbH, Berlin, Berlin
  - KPPK GmbH, Studienzentrum, Koblenz
  - Pneumologiezentrum Leipzig, Leipzig
  - Pneumologische Schwerpunktpraxis, 23558 Lübeck, Lübeck
- Netherlands (5):
  - Amphia Ziekenhuis, Breda
  - Zuyderland Medisch Centrum, Heerlen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Franciscus Gasthuis, Rotterdam
  - Gelre Ziekenhuis Zutphen, Zutphen
- Norway (4):
  - Frisk Utvikling Helse AS, Elverum
  - Hisøy Legesenter, Kolbjørnsvik
  - Lambertseter Legesenter, Oslo
  - Svelvik Legesenter, Svelvik

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://trials.boehringer-ingelheim.com/trial_results/ clinical_submission_documents.html to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link http://trials.boehringeringelheim.com/ to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://trials.boehringer-ingelheim.com

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A real-world, non-interventional study to assess the satisfaction of chronic obstructive pulmonary disease (COPD) patients with inhaler attributes and preferences for re-usable Respimat® Soft Mist Inhaler (SMI).
Pre-assignment Details: 262 patients were enrolled into the study, whereof 2 patients were enrolment failures as they did not meet eligibility criteria or received a disposable inhaler. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Respimat® SMI-experienced: Maintenance With Re-usable SMI: Chronic obstructive pulmonary disease (COPD) patients who had been on maintenance treatment with a re-usable Respimat Sof Mist Inhaler (SMI) product (Spiriva®, Striverdi®, or Spiolto®) at study entry. Patients were followed from the time of study entry (enrollment visit) for a period of approximately 4 to 6 weeks (study period).
- Respimat® SMI-experienced: Switching to Re-usable SMI: Chronic obstructive pulmonary disease (COPD) patients who had been on maintenance treatment with a disposable Respimat and who switched to a re-usable Respimat SMI at study entry. Patients were followed from the time of study entry (enrolment visit) for a period of approximately 4 to 6 weeks (study period).
- Respimat® SMI-naïve: Chronic obstructive pulmonary disease (COPD) patients who had not previously used a Respimat SMI product and had received their first prescription for a re-usable Respimat SMI product at study entry. Patients were followed from the time of study entry (enrolment visit) for a period of approximately 4 to 6 weeks (study period).
Period: Overall Study
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
Started | 133 | 71 | 56
Completed | 132 | 70 | 55
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Met exclusion criteria after study entry | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All enrolled patients who met all the eligibilty criteria of the study and who had received at least one dose of ther re-usable Respimat SMI product during the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve | Total
Number analyzed (Participants) | 133 | 70 | 56 | 259
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.1 (7.59) | 68.6 (8.58) | 68.7 (7.69) | 68.9 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 37 | 25 | 128
  Male | 67 | 33 | 31 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 131 | 66 | 56 | 253
  Unknown or Not Reported | 2 | 4 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 131 | 68 | 56 | 255
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Patient Satisfaction and Preference Questionnaire (PASAPQ) Score
Description: Total PASAPQ score is a measure of patient's satisfaction regarding the handling of the re-usable Respimat® SMI. The total score was the sum of the 13 items related to Performance and Convenience PASAPG domains (7 items for Performance domain: Q 1-5, 10-11, and 6 items for convenience domain: Q6-9, 12-13).
  Each PASAPQ item had response options ranging from 1 (very dissatisfied) to 7 (very satisfied). To calculate the total and domain score, the items within each domain were first summed and then transformed to a 0 (least) or 100 (most) point scale, with higher scores indicating greater satisfaction:
  Performance score = 100 *[(Q1+Q2 +Q3+ Q4+Q5+Q10+Q11)-7] /(49-7)
  Convenience score = 100 *[(Q6+ Q7+Q8+Q9+Q12+Q13)-6] / (42-6)
  Total score = 100 *[(Q1+Q2 +Q3+Q4+ Q5+Q6 + Q7+Q8+ Q9+Q10+Q11+Q12+Q13)-13] / (91-13)
Time Frame: At follow-up assessment, 4 to 6 weeks after baseline.
Population: Patients in the Full Analysis Set (FAS) who have available data for this endpoint.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
Number analyzed (Participants) | 131 | 69 | 55
Score on a scale | 84.26 [82.69 to 85.82] | 81.59 [78.71 to 84.47] | 83.24 [79.89 to 86.59]

2. Secondary Outcome: Total Performance PASAPQ Score for All Patients at Study End (Follow-up Assessment)
Description: The performance domain score of PASAPQ contained 7 items (Q 1-5 and 10-11), each item had response options ranging from 1 (very dissatisfied) to 7 (very satisfied). To calculate the domain score, the items were first summed and then transformed to a 0 (least) to 100 (most) point scale, with higher scores indicating greater satisfaction:
  Performance score = 100 * [(Q1+ Q2+Q3+Q4+Q5+Q10+Q11)-7] / (49-7)
Time Frame: At follow-up assessment, 4 to 6 weeks after baseline.
Population: Patients in the Full Analysis Set (FAS) who have available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
Number analyzed (Participants) | 131 | 69 | 55
Score on a scale | 84.70 (12.647) | 82.88 (14.938) | 82.38 (16.288)

3. Secondary Outcome: Total Convenience PASAPQ Score for All Patients at Study End (Follow-up Assessment)
Description: The convenience domain score of PASAPQ contained 6 items (Question 6-9 and 12-13), each item had response options ranging from 1 (very dissatisfied) to 7 (very satisfied). To calculate the domain score, the items were first summed and then transformed to a 0 (least) to 100 (most) point scale, with higher scores indicating greater satisfaction:
  Convenience score = 100 * [(Q6+Q7+Q8+Q9+Q12+Q13)-6] / (42-6)
Time Frame: At follow-up assessment, 4 to 6 weeks after baseline.
Population: Patients in the Full Analysis Set (FAS) who have available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
Number analyzed (Participants) | 131 | 69 | 55
Score on a scale | 83.74 (10.799) | 80.08 (15.075) | 84.24 (14.434)

4. Secondary Outcome: Overall Satisfaction Question With Inhaler for All Patients at Study End (Follow-up Assessment)
Description: The overall satisfaction score of the PASAPQ asked for the overall satisfaction with the device used in the study (Question 14), answered using a 7-point scale ranging from 1 (very dissatisfied) to 7 (very satisfied). Reported is the number of patients by category.
Time Frame: At follow-up assessment, 4 to 6 weeks after baseline.
Population: Patients in the Full Analysis Set (FAS) who have available data for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
Number analyzed (Participants) | 131 | 69 | 55
Participants
  Very dissatisfied | 0 | 1 | 1
  Dissatisfied | 2 | 0 | 0
  Somewhat dissatisfied | 1 | 2 | 1
  Neither satisfied nor dissatisfied | 3 | 3 | 1
  Somewhat satisfied | 7 | 4 | 3
  Satisfied | 69 | 36 | 25
  Very Satisified | 49 | 23 | 24

5. Secondary Outcome: Question on Willingness to Continue With Inhaler for All Patients at Study End (Follow-up Assessment)
Description: To assess the willingness to continue with inhaler, the following questions was asked: "How would you feel about continuing to use the inhaler?", using a value from 0-100, with zero indicating that the patient is not willing to continue using the inhaler and 100 indicating that the patient is definitely willing to continue using the inhaler.
Time Frame: At follow-up assessment, 4 to 6 weeks after baseline.
Population: Patients in the Full Analysis Set (FAS) who have available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
Number analyzed (Participants) | 131 | 69 | 54
Score on a scale | 89.1 (19.23) | 88.0 (19.29) | 84.1 (22.98)

6. Secondary Outcome: Questions on Ease of Handling of the Re-usable Respimat SMI for All Patients at Study End (Follow-up Assessment)
Description: 10 Questions regarding the Ease of Handling were asked, using a 7 point scale ranging from 1 (very dissatisfied) to 7 (very satisfied). Reported is the number of patients by answer category.
Time Frame: At follow-up assessment, 4 to 6 weeks after baseline.
Population: Full Analysis Set (FAS): All enrolled patients who met all the eligibility criteria of this study and who had received at least one dose of their re-usable Respimat SMI product during the study. Missing patients did not perform the Follow-up assesment or who did not perform the Ease of Handling assessment at Follow-Up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
Number analyzed (Participants) | 130 | 69 | 55
Participants
  Q1: How satisfied are you with the ease of removing the clear base?: Very dissatisfied | 0 | 3 | 1
  Q1: How satisfied are you with the ease of removing the clear base?: Dissatisfied | 4 | 2 | 0
  Q1: How satisfied are you with the ease of removing the clear base?: Somewhat dissatisfied | 3 | 5 | 0
  Q1: How satisfied are you with the ease of removing the clear base?: Neither satisfied nor dissatisfied | 5 | 5 | 2
  Q1: How satisfied are you with the ease of removing the clear base?: Somewhat satisfied | 5 | 4 | 5
  Q1: How satisfied are you with the ease of removing the clear base?: Satisfied | 64 | 29 | 26
  Q1: How satisfied are you with the ease of removing the clear base?: Very satisfied | 49 | 21 | 21
  Q1: How satisfied are you with the ease of removing the clear base?: Not applicable | 0 | 0 | 0
  Q2: How satisfied are you with the grip of the cartridge?: number analyzed (Participants) | 130 | 69 | 54
  Q2: How satisfied are you with the grip of the cartridge?: Very dissatisfied | 0 | 2 | 0
  Q2: How satisfied are you with the grip of the cartridge?: Dissatisfied | 3 | 2 | 0
  Q2: How satisfied are you with the grip of the cartridge?: Somewhat dissatisfied | 2 | 2 | 0
  Q2: How satisfied are you with the grip of the cartridge?: Neither satisfied nor dissatisfied | 2 | 1 | 2
  Q2: How satisfied are you with the grip of the cartridge?: Somewhat satisfied | 6 | 1 | 4
  Q2: How satisfied are you with the grip of the cartridge?: Satisfied | 66 | 38 | 31
  Q2: How satisfied are you with the grip of the cartridge?: Very satisfied | 51 | 23 | 17
  Q2: How satisfied are you with the grip of the cartridge?: Not applicable | 0 | 0 | 0
  Q3: How satisfied are you with inserting a new cartridge?: Very dissatisfied | 0 | 3 | 0
  Q3: How satisfied are you with inserting a new cartridge?: Dissatisfied | 7 | 3 | 0
  Q3: How satisfied are you with inserting a new cartridge?: Somewhat dissatisfied | 5 | 6 | 2
  Q3: How satisfied are you with inserting a new cartridge?: Neither satisfied nor dissatisfied | 4 | 3 | 4
  Q3: How satisfied are you with inserting a new cartridge?: Somewhat satisfied | 10 | 6 | 5
  Q3: How satisfied are you with inserting a new cartridge?: Satisfied | 57 | 31 | 30
  Q3: How satisfied are you with inserting a new cartridge?: Very satisfied | 47 | 17 | 14
  Q3: How satisfied are you with inserting a new cartridge?: Not applicable | 0 | 0 | 0
  Q4: How satisfied are you with the readability of the dose indicator?: number analyzed (Participants) | 130 | 68 | 55
  Q4: How satisfied are you with the readability of the dose indicator?: Very dissatisfied | 1 | 3 | 1
  Q4: How satisfied are you with the readability of the dose indicator?: Dissatisfied | 4 | 0 | 0
  Q4: How satisfied are you with the readability of the dose indicator?: Somewhat dissatisfied | 4 | 1 | 0
  Q4: How satisfied are you with the readability of the dose indicator?: Neither satisfied nor dissatisfied | 1 | 0 | 1
  Q4: How satisfied are you with the readability of the dose indicator?: Somewhat satisfied | 5 | 2 | 4
  Q4: How satisfied are you with the readability of the dose indicator?: Satisfied | 62 | 27 | 34
  Q4: How satisfied are you with the readability of the dose indicator?: Very satisfied | 53 | 35 | 15
  Q4: How satisfied are you with the readability of the dose indicator?: Not applicable | 0 | 0 | 0
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Very dissatisfied | 0 | 1 | 0
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Dissatisfied | 2 | 1 | 0
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Somewhat dissatisfied | 3 | 2 | 2
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Neither satisfied nor dissatisfied | 3 | 0 | 4
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Somewhat satisfied | 5 | 2 | 1
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Satisfied | 65 | 35 | 33
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Very satisfied | 52 | 28 | 15
  Q5: How satisfied are you with recognising when you need to replace the cartridge?: Not applicable | 0 | 0 | 0
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: number analyzed (Participants) | 129 | 68 | 55
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Very dissatisfied | 0 | 1 | 0
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Dissatisfied | 4 | 4 | 0
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Somewhat dissatisfied | 1 | 3 | 2
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Neither satisfied nor dissatisfied | 6 | 5 | 2
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Somewhat satisfied | 10 | 5 | 5
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Satisfied | 65 | 31 | 33
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Very satisfied | 43 | 19 | 13
  Q6: How satisfied are you with automatic detachment of the clear base when the cartridge is empty?: Not applicable | 0 | 0 | 0
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: number analyzed (Participants) | 129 | 68 | 55
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Very dissatisfied | 0 | 1 | 0
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Dissatisfied | 3 | 2 | 0
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Somewhat dissatisfied | 4 | 7 | 0
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Neither satisfied nor dissatisfied | 7 | 6 | 6
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Somewhat satisfied | 5 | 2 | 2
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Satisfied | 69 | 35 | 30
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Very satisfied | 41 | 15 | 17
  Q7: How satisfied are you with automatic return to start-use position when replacing the clear base?: Not applicable | 0 | 0 | 0
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Very dissatisfied | 0 | 3 | 0
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Dissatisfied | 2 | 0 | 0
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Somewhat dissatisfied | 2 | 1 | 0
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Neither satisfied nor dissatisfied | 2 | 4 | 3
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Somewhat satisfied | 1 | 1 | 3
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Satisfied | 69 | 35 | 27
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Very satisfied | 54 | 25 | 22
  Q8: How satisfied are you with the overall ease of handling the inhaler?: Not applicable | 0 | 0 | 0
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Very dissatisfied | 2 | 2 | 0
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Dissatisfied | 1 | 1 | 0
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Somewhat dissatisfied | 0 | 2 | 1
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Neither satisfied nor dissatisfied | 7 | 3 | 1
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Somewhat satisfied | 4 | 2 | 5
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Satisfied | 49 | 26 | 26
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Very satisfied | 67 | 33 | 22
  Q9: How satisfied are you with the sustainability concept of the inhaler, due to re-use ability?: Not applicable | 0 | 0 | 0
  Q10: How satisfied are you with recognising when to replace the inhaler?: number analyzed (Participants) | 129 | 69 | 55
  Q10: How satisfied are you with recognising when to replace the inhaler?: Very dissatisfied | 1 | 1 | 0
  Q10: How satisfied are you with recognising when to replace the inhaler?: Dissatisfied | 3 | 2 | 0
  Q10: How satisfied are you with recognising when to replace the inhaler?: Somewhat dissatisfied | 1 | 0 | 0
  Q10: How satisfied are you with recognising when to replace the inhaler?: Neither satisfied nor dissatisfied | 4 | 1 | 2
  Q10: How satisfied are you with recognising when to replace the inhaler?: Somewhat satisfied | 7 | 2 | 2
  Q10: How satisfied are you with recognising when to replace the inhaler?: Satisfied | 54 | 39 | 26
  Q10: How satisfied are you with recognising when to replace the inhaler?: Very satisfied | 56 | 20 | 22
  Q10: How satisfied are you with recognising when to replace the inhaler?: Not applicable | 3 | 4 | 3

7. Secondary Outcome: Difference in the Mean Total PASAPQ Score Between Study Entry and Study End in Respimat SMI-experienced Patients Who Switched From a Disposable to a Re-usable Respimat SMI Product
Description: Difference in the mean Total PASAPQ score between study entry (baseline visit) and at study end (follow-up assessment) in Respimat SMI-experienced patients who switched from a disposable to a re-usable Respimat SMI product at study entry.
  The total score was the sum of the 13 items related to Performance and Convenience PASAPG domains (7 items for Performance domain: Q 1-5, 10-11, and 6 items for convenience domain: Q6-9, 12-13).
  Each PASAPQ item had response options ranging from 1 (very dissatisfied) to 7 (very satisfied). To calculate the total and domain score, the items within each domain were first summed and then transformed to a 0 (least) or 100 (most) point scale, with higher scores indicating greater satisfaction.
Time Frame: At study entry (baseline) and at study end (4 to 6 weeks after baseline).
Population: FAS: Respimat SMI-experience patients who switched from a disposable to a re-usable Respimat SMI product at study entry and with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Respimat® SMI-experienced: Switching to Re-usable SMI
Number analyzed (Participants) | 68
Score on a scale | 1.10 (10.034)

8. Secondary Outcome: Number of Patients With Preference for Re-usable or Disposable Respimat SMI at Study End in Respimat SMI-experienced Patients Who Switched From a Disposable to a Re-usable Respimat SMI Product
Description: Number of patients with preference for re-usable or disposable Respimat SMI at study end (follow-up assessment), in Respimat SMI-experienced patients who switched from a disposable to a re-usable Respimat SMI product at study entry. To assess the preference for inhaler, following question was asked: "Comparing the re-usable with disposable inhaler, which inhaler do you prefer to use?"
Time Frame: At follow-up assessment, 4 to 6 weeks after baseline.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Respimat SMI-experienced Patients Switching to a Re-usable Respimat SMI at Study Entry: Respimat SMI-experienced patients switching to a re-usable Respimat SMI at study entry.
Arm/Group | Respimat SMI-experienced Patients Switching to a Re-usable Respimat SMI at Study Entry
Number analyzed (Participants) | 68
Participants
  Re-usable inhaler | 57
  Disposable inhaler | 8
  No preference | 3

ADVERSE EVENTS:
Time Frame: From study entry until end of study, up to 6 weeks.
Description: Full Analysis Set (FAS): All enrolled patients who met all the eligibility criteria of the study and who had received at least one dose of ther re-usable Respimat SMI product during the study period.
Arm/Group | Respimat® SMI-experienced: Maintenance With Re-usable SMI | Respimat® SMI-experienced: Switching to Re-usable SMI | Respimat® SMI-naïve
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/70 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/70 | 0/56
Other Adverse Events (participants affected / at risk) | 0/133 | 0/70 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review Prior to any Submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI´s intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT04011735/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT04011735/SAP_001.pdf